CLINICAL TRIAL: NCT06578247
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Trial Of Quizartinib Administered in Combination With Induction and Consolidation Chemotherapy and Administered as Maintenance Therapy in Adult Patients With Newly Diagnosed FLT3-ITD Negative Acute Myeloid Leukemia
Brief Title: Quizartinib or Placebo Plus Chemotherapy in Newly Diagnosed Patients With FLT3-ITD Negative AML
Acronym: QuANTUM-WILD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC220-168; 2023-507936-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-14; First posted 2024-08-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Leukemia
Keywords: acute myeloid leukemia; quizartinib; FLT3; FLT3-ITD; Chemotherapy; FLT3-WT
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — quizartinib; Drug Therapy; Cytarabine; Daunorubicin; Idarubicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study has a double-blind design. Neither the participants nor any of the investigators, Sponsor, Independent Review Committee (IRC) or contract research organizations (CROs) will be aware of the treatments received. An independent biostatistician, not otherwise part of the Sponsor trial team, will generate the randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Quizartinib + Chemotherapy (Experimental): Participants will receive quizartinib at 60 mg/day orally once daily for 14 days starting after the completion of chemotherapy in Induction and Consolidation Phase. In the Maintenance Phase, participants will receive quizartinib at 60 mg/day orally once daily for up to 36 cycles (28-day cycle)
  Interventions: Drug: Quizartinib; Drug: Chemotherapy
- Arm B: Placebo + Chemotherapy (Placebo Comparator): Participants will receive placebo at 60 mg/day orally once daily for 14 days starting after the completion of chemotherapy in Induction and Consolidation Phase. In the Maintenance Phase, participants will receive placebo at 60 mg/day orally once daily for up to 36 cycles (28-day cycle)
  Interventions: Drug: Placebo; Drug: Chemotherapy
- Arm C: Quizartinib + Chemotherapy then Placebo Maintenance (Experimental): Participants will receive quizartinib at 60 mg/day orally once daily for 14 days starting after the completion of chemotherapy in Induction and Consolidation Phase. In the Maintenance Phase, participants will receive placebo at 60 mg/day orally once daily for up to 36 cycles (28-day cycle)
  Interventions: Drug: Quizartinib; Drug: Placebo; Drug: Chemotherapy

INTERVENTIONS:
Drug: Quizartinib — Participants will receive quizartinib at 60 mg/day orally once daily
  Other Names: Test Product
  Arms: Arm A: Quizartinib + Chemotherapy; Arm C: Quizartinib + Chemotherapy then Placebo Maintenance
Drug: Placebo — Participants will receive placebo at 60 mg/day orally once daily
  Other Names: Placebo Control
  Arms: Arm B: Placebo + Chemotherapy; Arm C: Quizartinib + Chemotherapy then Placebo Maintenance
Drug: Chemotherapy — Participants will receive commercially available cytarabine (cytosine arabinoside) and anthracycline (daunorubicin or idarubicin).
  Other Names: Cytarabine, Daunorubicin or Idarubicin; Standard Chemotherapy

SUMMARY:
This study will compare the effects of Quizartinib versus placebo in combination with chemotherapy in participants with newly diagnosed FMS-like tyrosine kinase 3 (FLT3)-internal tandem duplication (ITD) negative acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This is a clinical trial to compare the effect of quizartinib versus placebo (administered with standard induction and consolidation chemotherapy, then administered as maintenance therapy for up to 36 cycles) on the primary endpoint of overall survival (OS) in adult patients with newly diagnosed FMS-like tyrosine kinase 3 (FLT3)-internal tandem duplication (ITD) negative acute myeloid leukemia (AML). Participants will be tested for FLT3-ITD mutation status in a central laboratory using a validated assay.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must be competent and able to comprehend, sign, and date an Ethics Committee (EC)- or Institutional Review Board (IRB)-approved ICF before performance of any trial-specific procedures or tests.
2. ≥18 years or the minimum legal adult age (whichever is greater) and ≤70 years (at Screening).
3. Newly diagnosed, morphologically documented primary AML based on the World Health Organization (WHO) 2016 classification (at Screening)
4. Eastern Cooperative Oncology Group (ECOG) performance status (at the time the participant signs their ICF) of 0-2.
5. Participant is a candidate for standard "7+3" induction chemotherapy regimen as specified in the protocol per investigator assessment

Key Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL), French-American-British classification M3 or WHO classification of APL with translocation, t(15;17)(q22;q12), or BCR-ABL positive leukemia (ie, chronic myelogenous leukemia in blast crisis); participants who undergo diagnostic workup for APL and treatment with all-trans retinoic acid (ATRA), but who are found not to have APL, are eligible (treatment with ATRA must be discontinued before starting induction chemotherapy).
2. Diagnosis of AML secondary to prior chemotherapy or radiotherapy.
3. Diagnosis of AML with known antecedent myelodysplastic syndrome (MDS) or a myeloproliferative neoplasm (MPN) or MDS/MPNs including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), juvenile myelomonocytic leukemia (JMML) and others.
4. Participants with newly diagnosed AML with FLT3-ITD mutations (FLT3-ITD [+]) present at ≥5% VAF (or ≥0.05 SR) based on a validated FLT3 mutation assay.
5. Prior treatment for AML, except for the following allowances prior to Day 1 of chemotherapy:

   1. Leukapheresis;
   2. Treatment for hyperleukocytosis with hydroxyurea;
   3. Cranial radiotherapy for central nervous system (CNS) leukostasis;
   4. Prophylactic intrathecal chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2030-06-26 (Estimated); Study Completion 2030-06-26 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (Arm A vs Arm B) | Date of first patient randomized to the target number of deaths reached, up to approximately 42 months
  Overall survival (OS) is defined as the time from randomization until death from any cause.

SECONDARY OUTCOMES:
Event-free survival (Arm A vs. Arm B) | Date of randomization up to approximately 42 months
  Event-free survival (EFS) is defined as time from randomization to date of failure to achieve CR at end of induction, relapse after CR, or death due to any cause, whichever occurs first
Duration of complete response (Arm A vs. Arm B) | Date of randomization up to approximately 42 months
  Duration of complete response (DoCR) is defined as time from the first documented CR until documented relapse or death due to any cause, whichever comes first. As assessed by Independent Review Committee.
Relapse-free survival (Arm A vs. Arm B) | Date of randomization up to approximately 42 months
  Relapse-free survival (RFS) is defined as time from randomization, for participants who achieve CR in the Induction Phase, until relapse or death due to any cause, whichever comes first. As assessed by Independent Review Committee .
Complete remission rate (Arm A vs. Arm B) | At end of Induction Phase, up to approximately 120 days
  Complete remission rate (CR) is defined as proportion of of participants who achieved a CR. As assessed by Independent Review Committee.
Complete remission rate with minimal or measurable residual disease (Arm A vs. Arm B) | At end of Induction Phase (Cycle 2 or Cycles 1 and 2), up to approximately 120 days
  Proportion of participants achieving CR with minimal or measurable residual disease (MRD) negativity. As assessed by Independent Review Committee.
Number of Participants With Treatment-emergent Adverse Events (Arm A vs. Arm B) | Date of first dose up to 30 days after last dose, up to approximately 42 months
  Treatment-emergent adverse events (TEAE) are defined as those AEs with start or worsening date during the on-treatment period (from the first dose date of quizartinib/placebo to 30 days after the last dose date of quizartinib/placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (286):
- United States (51):
  - City of Hope Phoenix, Goodyear, Arizona
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - David Geffen School of Medicine, Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - Ucsf - School of Medicine, San Francisco, California
  - Stanford University School of Medicine- Parent, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Florida Hospital Cancer Institute - Kissimmee, Kissimmee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Robert H Lurie Comprehensive Cancer Center Northwestern University, Chicago, Illinois
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Medical Center - New Orleans, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Medical School - Twin Cities Campus, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Thomas Jefferson Univ Hosp, Haddonfield, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - Main, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - Main, New York, New York
  - Upstate University Hospital, Syracuse, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke Cancer Institute - Sarcoma Research, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Ohio Health Marion Area Physicians, Columbus, Ohio
  - Peggy & Charles Stephenson Oklahoma Cancer Ctr, Oklahoma City, Oklahoma
  - Oregon Health & Science University (Ohsu), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Upmc Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Tristar Bone Marrow Transplant, Nashville, Tennessee
  - South Austin Medical Center, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Uva Health System, Charlottesville, Virginia
  - Virginia Commonwealth University (Vcu) Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (11):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre (Fmc), Bedford Park
  - Box Hill Hospital, Box Hill
  - Concord Repatriation General Hospital, Concord
  - St Vincent'S Hospital Melbourne, Darlinghurst
  - Townsville University Hospital, Douglas
  - Liverpool Hospital, Liverpool
  - The Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital, Perth
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Ordensklinikum Linz Gmbh - Elisabethinen, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Hanusch Krankenhaus Der Wgkk Wien, Vienna
- Belgium (6):
  - Institut Jules Bordet, Anderlecht
  - ZNA, Antwerp
  - Az Sint-Jan, Bruges
  - Uz Leuven, Leuven
  - Chu of Liège, Liège
  - AZ DELTA, Roeselare
- Brazil (24):
  - Cetus Hospital Dia Oncologia, Belo Horizonte
  - Unesp - Faculdade de Medicina Da Universidade Estadual Paulista - Campus Botucatu, Botucatu
  - Centro de Hematologia E Hemoterapia - Hemocentro de Campinas - Unicamp, Campinas
  - Centro de Hematologia e Hemoterapia - Hemocentro de Campinas - UNICAMP, Campinas
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - Hospital Erasto Gaertner - Liga Paranaense de Combate Ao Că'Ncer, Curitiba
  - Cepon - Centro De Pesquisas Oncolagicas de Santa Catarina, Florianópolis
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - Hc-Ufg - Hospital Das Clă Nicas Da Universidade Federal de Goiă S, Goiânia
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Fundaã§Ã£O Doutor Amaral Carvalho, Jaú
  - Hospital de Clínicas de Passo Fundo, Passo Fundo
  - Hospital de Clă Nicas de Passo Fundo, Passo Fundo
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Clă Nicas de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - INCA - Instituto Nacional de Cancer, Rio de Janeiro
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, Sao Jose Rio Preto
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
  - Hospital Beneficencia Portuguesa da Sao Paulo, São Paulo
  - Hospital Nove de Julho, São Paulo
  - Sírio-Libanês Brasilia-Centro de Oncologia-Asa Sul, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo Octavio Frias de Oliveira, SĂŁo Paulo
- Bulgaria (6):
  - Umhat 'Dr. Georgi Stranski', Ead, Pleven
  - Umhat 'Sv. Georgi', Ead, Plovdiv
  - Umhat Â Sv. Ivan Rilskiâ , Ead, Sofia
  - Military Medical Academy - Mhat - Sofia, Sofia
  - 'Shathd' Ead Sofia, Sofia
  - Umhat Prof. Dr. Stoyan Kirkovich Ad, Stara Zagora
- Canada (5):
  - London Health Sciences Centre, London
  - McGill University - Dept. Oncology Clinical Research Program, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - Saskatoon Cancer Centre, Saskatoon
  - Princess Margaret Cancer Center, Toronto
- China (27):
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central South University, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Sun Yat-Sen University, Cancer Center, Guangzhou
  - Guangdong Provincial People'S Hospital, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhong Da Hospital, Southeast University, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Shanghai Tongren Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shengyang
  - Shenzhen Second People'S Hospital, Shenzhen
  - The Second Hospital of Hebei Medicical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematology and Hospital of Blood Disease, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuxi People'S Hospital, Wuxi
  - The First Affiliated Hospital of Xiâ An Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- Croatia (3):
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centar Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
- Czechia (6):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Plzen, Pilsen
  - Fakultni Nemocnice Ostrava, Poruba
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Ustav Hematologie A Krevni Transfuze, Prague
- France (17):
  - Chu Angers - Hă"Pital Hă"Tel Dieu, Angers
  - Chu de Caen, Caen
  - Chu de Grenoble - Hospital Albert Michallon, La Tronche
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hopital Claude Huriez - Chru Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hopital de La Conception - Aphm, Marseille
  - Chu de Nantes - Hotel Dieu, Nantes
  - CHU Nice - Hôpital de l'Archet 1, Nice
  - Hospital Saint-Louis, Paris
  - Chu de Bordeaux - Hă"Pital Haut-Lă Vă Que, Pessac
  - Centre Hospitalier Lyon Sud, Pierre BĂŠnite
  - Chu Rennes - Hopital Pontchaillou, Rennes
  - Chu Amiens - Hopital Sud, Salouël
  - Institut de Cancă Rologie de Strasbourg Europe - Icans, Strasbourg
  - Institut Universitaire Du Cancer de Toulouse- Iuct-O, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Klinikum Aschaffenburg-Alzenau, Alzenau in Unterfranken
  - Charité Campus Virchow-Klinikum, Berlin
  - Staedtisches Klinikum Braunschweig Ggmbh, Braunschweig
  - Universitaetsklinikum Carl Gustav Carus Tu Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Krh Klinikum Siloah, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universită"Tsklinikum Leipzig Klinik Fă R Hă"Matologie Internistische Onkologie Hă"Mostaseol, Leipzig
  - Universitaetsklinikum Muenster, Münster
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong (Cuhk), Shatin
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Italy (14):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico Di Bari, Bari
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia (Presidio Spedali Civili), Brescia
  - Irccs Istituto Scientifico Romagnolo Per Lo Studio Dei Tumori 'Dino Amadori' - Irst, Meldola
  - Ospedale San Raffaele, Milan
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Ospedale Maggiore Di Novara, Novara
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Istituto Clinico Humanitas, Rozzano
  - Irccs Ospedale Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliero-Universitaria Cittă Della Salute E Della Scienza Di Torino, Torino
  - Ospedale Mauriziano Umberto I, Torino
  - Asst Dei Sette Laghi Ospedale Di Circolo E Fondazione Macchi Varese, Varese
- Japan (18):
  - Akita University Hospital, Akita
  - Aomori Prefetural Central Hospital, Aomori
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō City
  - Chiba Aoba Municipal Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Chugoku Central Hospital, Fukuyama
  - Gifu Municipal Hospital, Gifu
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu
  - Tesshokai Kameda General Hospital, Kamogawa-shi
  - Kanazawa University Hospital, Kanazawa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Saiseikai Maebashi Hospital, Maebashi
  - Ehime Prefectural Central Hospital, Matsuyama
  - Nagoya University Hospital, Nagoya
  - Japan RED CROSS OSAKA HOSPITAL, Osakar
  - Hokkaido University Hospital, Sapporo
  - Sapporo Hokuyu Hospital, Sapporo
  - Tenri Hospital, Tenri
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, TromsĂ¸
- Poland (4):
  - Klinika Hematoonkologii I Transplantacji Szpiku, Lublin
  - Spzoz Msw Zwarmiĺsko-Mazurskimcen.Onko.Wolsztynie, Olsztyn
  - Wojewodzki Szpital Zespolony Im. L. Rydygiera W Toruniu, Torun
  - Instytut Hematologii I Transfuzjologii, Warsaw
- Portugal (2):
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Portugues De Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (5):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Municipal Filantropia Craiova, Craiova
- Serbia (3):
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center Nis, Niš
- Singapore (2):
  - National University Hospital, Singapore
  - Curie Oncology Pte Ltd, Singapore
- South Korea (17):
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary'S Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (25):
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Ico Badalona - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario De Burgos, Burgos
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas
  - Clinica Universidad de Navarra, Madrid
  - Md Anderson Cancer Centre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gasteborg
  - Skă Nes Universitetssjukhus, Lund, Lund
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Luzerner Kantonsspital - Luzern, Lazern 16
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospitalx, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - King'S College Hospital, London
  - Hammersmith Hospital, London
  - Maidstone Hospital, Maidstone
  - Manchester Royal Infirmary, Manchester
  - Churchill Hospital, Oxford
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/